CLINICAL TRIAL: NCT02826525
Title: Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD4076 Following Multiple Ascending Dose Administration to T2DM Subjects With Non-Alcoholic Fatty Liver Disease
Brief Title: AZD4076 in Type 2 Diabetic Subjects With Non-Alcoholic Fatty Liver Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D5590C00002
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: T2DM With NAFLD
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Subjects in this arm will receive AZD4076
  Interventions: Drug: AZD4076
- Control (Placebo Comparator): Subjects in this arm will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4076 — Investigational product
  Other Names: Study drug
  Arms: Treatment
Drug: Placebo — Control
  Other Names: Control
  Arms: Control

SUMMARY:
This is a phase I/IIa, randomized, single-blind, placebo-controlled, multiple-ascending dose study conducted at a single site. The study plans to include up to approximately 46 evaluable subjects with Type 2 Diabetes Mellitus (HbA1c 7-11%) and Non-Alcoholic Fatty Liver disease (liver fat content > = 8%) on metformin monotherapy.

Three initial cohorts are planned:

* Cohort 1: 6 subjects receiving AZD4076 and 4 subjects receiving placebo
* Cohort 2: 12 subjects receiving AZD4076 and 10 subjects receiving placebo
* Cohort 3: 10 subjects receiving AZD4076 and 10 subjects receiving placebo, with the possibility to add additional subjects if drop-out rates are higher than expected

Pending review by SRC, an additional 2 cohorts, each consisting of 18 evaluable subjects may be included in the study.

The primary objectives of this clinical trial are to investigate the safety and tolerability of AZD4076 following subcutaneous administration of multiple ascending doses; to assess the effect of AZD4076 on whole body insulin sensitivity using hyperinsulinemic euglycemic clamp with tracer technique; and to assess the effect of AZD4076 on liver fat content using magnetic resonance imaging. Secondary objectives of this trial are to characterize multiple dose PK of AZD4076 and its longmer and shortmer metabolites and assess the time required to reach steady state and the degree of accumulation; to assess the efficacy of AZD4076 on 24-hour glucose; and to assess the effect of AZD4076 on homeostatic model assessment insulin resistant (HOMA-IR) and Matsuda index.

DETAILED DESCRIPTION:
This is a phase I/IIa, randomized, single-blind, placebo-controlled, multiple-ascending dose study conducted at a single site. The study plans to include up to approximately 46 evaluable subjects with Type 2 Diabetes Mellitus (HbA1c 7-11%) and Non-Alcoholic Fatty Liver disease (liver fat content > = 8%) on metformin monotherapy

Three initial cohorts are planned:

* Cohort 1: 6 subjects receiving AZD4076 and 4 subjects receiving placebo
* Cohort 2: 12 subjects receiving AZD4076 and 10 subjects receiving placebo
* Cohort 3: 10 subjects receiving AZD4076 and 10 subjects receiving placebo, with the possibility to add additional subjects if drop-out rates are higher than expected.

Pending review by SRC, an additional 2 cohorts, each consisting of 18 evaluable subjects may be included in the study.

The planned study consists of a screening visit, followed by 12 subsequent study visits. There will be a total of three residential periods: (1) Loading phase of the treatment (visit 2, days -4 to 14), (2) maintenance phase of treatment (visit 6, days 42-43), and (3) 8 weeks post-first dose of study drug (visit 9, days 53-56). Dosing of study drug will take place on days 1, 3, 5, 7, and 9 in the loading phase; and on days 14, 21, 28, 35, and 42 during the maintenance phase. Following the maintenance phase, subjects will have four follow-up visits.

Study Objectives:

The primary objectives of this clinical trial are to investigate the safety and tolerability of AZD4076 following subcutaneous administration of multiple ascending doses; to assess the effect of AZD4076 on whole body insulin sensitivity using hyperinsulinemic euglycemic clamp with tracer technique; and to assess the effect of AZD4076 on liver fat content using magnetic resonance imaging. Secondary objectives of this trial are to characterize multiple dose PK of AZD4076 and its longmer and shortmer metabolites and assess the time required to reach steady state and the degree of accumulation; to assess the efficacy of AZD4076 on 24-hour glucose; and to assess the effect of AZD4076 on homeostatic model assessment insulin resistant (HOMA-IR) and Matsuda index.

Study Population:

Subjects participating in this study are adult males and females of non-child bearing potential, who are 18-70 years of age, body mass index 23-40 kg/m2, diagnosed with T2DM who are inadequately controlled (HbA1C 7-11%) on a stable metformin regimen, and who have hepatic steatosis (defined as liver fat content of >=8% per MRI).

Duration of treatment:

The screening visit will occur within 42 days prior to the administration of the study drug. Total length of the treatment period is 6 weeks. The treatment period is divided in two phases: the loading phase, in which participants will receive the study drug every other day for 9 days (Days 1, 3, 5 , 7 and 9); thereafter subjects will enter the maintenance phase, where dosing will occur once weekly for four weeks (Days 14, 21, 28, 35 and 42). To ensure safety, subjects will be followed for approximately 5 months post the last dose of study drug.

Investigational product, dosage and mode of administration:

The study will utilize two study drugs: AZD4076 and placebo. Both drugs will be administered subcutaneously in the abdomen.

Safety analysis:

The key outcomes for the safety analyses are: adverse events, vital signs, safety laboratory parameters, ECGs, telemetry; and structured neurological and physical examination, as well as injection site assessment. Pharmacodynamic parameters will be derived from data generated from the clamp procedure, MRI, HOMA, OGTT and 24-hour glucose AUC. For pharmacokinetic parameters, plasma and urine concentrations of AZD4076 and its metabolites will be measured

ELIGIBILITY:
Inclusion criteria

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Males or females of non-child bearing potential.
3. Age 18-70 years with suitable veins for cannulation or repeated venipuncture.
4. BMI 23-40 kg/m2 inclusive.
5. Diagnosed T2D (HbA1c 7-11%) treated with a stable dose of metformin for at least one month prior to screening.
6. Hepatic steatosis of ≥8%.

Exclusion criteria

1. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
2. History or presence of hepatic or renal disease (with the exception of hepatic steatosis).
3. Presence of acute proliferative retinopathy or maculopathy, severe gastroparesis, and/or severe neuropathy, in particular autonomic neuropathy.
4. Clinically significant cardiovascular event within the last 6 months prior to screening.
5. History or presence of significant neurological or psychiatric disease/mental illness (as assessed using the C-SSRS).
6. History of malignancy within the last 5 years, excluding successful treatment of basal cell skin carcinoma or in situ carcinoma of cervix.
7. Suspicion of or known Gilbert's syndrome.
8. Supine systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 95 mmHg confirmed in the screening period.
9. Changes in any current medication (initiation, dose change or cessation) that may impact the study readouts (as judged by the Investigator) within three months prior to MRI assessment of steatosis screening. The criterion does not apply to medication prescribed for occasional use.

10 Treatment with antidiabetics (except for metformin) during the last three months prior to screening or treatment with sulfonylurea (SU) drugs within the 4 weeks prior to screening.

11. Used or plan to use drugs that cause weight loss, participating in, or have participated in weight loss program within the last 3 months.

12. Use of anabolic steroids and systemic treatment with glucosteroids within three months prior to screening. Intra articular, topical, and inhaled steroids are permissible.

13. Any confirmed clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the Investigator.

14. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV).

15. Confirmed serum creatinine greater than the ULN. 16. A confirmed eGFR <60 calculated according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.

17. Confirmed platelet count outside the normal range. 18. Confirmed ALT or AST greater than 1.5x ULN. 19. Confirmed total bilirubin greater than ULN 20. Any clinically significant abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG, as considered by the investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead, or left ventricular hypertrophy.

21. Prolonged QTcF > 450 ms for males and > 470 ms for females or family history of long QT syndrome.

22. PR(PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation.

23. PR (PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree AV block, or AV dissociation.

24. Persistent or intermittent complete bundle branch block (BBB) with QRS > 120 ms.

25. Known or suspected history of drug abuse within the past 5 years, as judged by the Investigator.

26. Smokes >10 cigarettes/day and unable to comply with the nicotine restriction during the study.

27. History of alcohol abuse or excessive intake of alcohol. Definition of excessive intake: an average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits.

28. Positive screen for drugs of abuse at screening or admission to the unit or positive screen for alcohol at screening or on admission to the unit prior to the first administration of IMP.

29. History of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4076.

30. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea), as judged by the Investigator.

31. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.

32. Plasma donation within one month of screening or any blood donation/blood loss > 500 mL during the 56 days prior to screening.

33. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within one month of the administration of IMP in this study. The period of exclusion begins one month after the final dose or one month after the last visit whichever is the longest.

34. Use of implants or devices that are incompatible with the MRI procedure. 35. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

36. Involvement of any Astra Zeneca, PROFIL INSTITUTE or study site employee or their close relatives.

37. Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.

38. Subjects not willing to comply with the dietary requirements in the study as judged by the Investigator.

39. Subjects who cannot communicate reliably with the Investigator or designee. 40. Previous bone marrow transplant. 41. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of AZD4076 by assessing the number of participants with adverse events | From screening until 26 weeks post first dose
  To assess the safety and tolerability of multiple ascending doses of AZD4076
The safety and tolerability of AZD4076 by assessment of blood pressure | From screening until 26 weeks post first dose
  To assess the safety and tolerability of multiple ascending doses of AZD4076
The safety and tolerability of AZD4076 by assessment of pulse | From screening until 26 weeks post first dose
  To assess the safety and tolerability of multiple ascending doses of AZD4076
The safety and tolerability of AZD4076 by assessment of oral temperature | From day -2 until day 42
  To assess the safety and tolerability of multiple ascending doses of AZD4076
The safety and tolerability of AZD4076 by assessment of electrocardiogram readings | From screening until 26 weeks post first dose
  To assess the safety and tolerability of multiple ascending doses of AZD4076
The safety and tolerability of AZD4076 by assessment of digital electrocardiogram readings | From predose until 24 hours post-dose on days 1 and 42
  To assess the safety and tolerability of multiple ascending doses of AZD4076
The safety and tolerability AZD4076 by assessment of physical examination | From screening until 26 weeks post first dose
  Percentage of patients with abnormal physical examination
The safety and tolerability of AZD4076 by assessing the injection site | From day 1 until day 42
  Percentage of patients with dermatological adverse events
The safety and tolerability of AZD4076 by assessing the number of adverse events | From screening until 26 weeks post first dose
  To assess the safety and tolerability of multiple ascending doses of AZD4076
The safety and tolerability of AZD4076 by assessing hematology | From screening until 26 weeks post first dose
  To assess the safety and tolerability of multiple ascending doses of AZD4076
The safety and tolerability of AZD4076 by assessing clinical chemistry | From screening until 26 weeks post first dose
  Percentage of patients with clinically significant changes in laboratory tests.
The safety and tolerability of AZD4076 by assessing urinalysis | From screening until 26 weeks post-first dose
  To assess the safety and tolerability of multiple ascending doses of AZD4076
Glucose infusion rate at hyperinsulinemic clamp | Day -1 and 56 days post first dose
  To assess the effect of AZD4076 on whole body insulin sensitivity using hyperinsulinemic euglycemic clamp with tracer technique
Reduction in liver fat content (%) per MRI | Screening and 54 days post first dose
  To assess the effect of AZD4076 on liver fat content using magnetic resonance imaging

SECONDARY OUTCOMES:
24 hour glucose area under the curve | Day -2 and day 55
  To assess the effect of AZD4076 on 24-hour glucose.
HOMA-IR | Day -2 and day 55
  To assess the effect of AZD4076 on homeostatic model assessment insulin resistant (HOMA-IR)
Fasting Endogenous Glucose Production | Day -1 and day 56
  To assess the effect of AZD4076 on endogenous glucose production (EGP).
AUCt of AZD4076 and longmer and shortmer metabolites | Dosing day 1 and day 42
  To characterize pharmacokinetics of AZD4076 by area under the curve to time
Matsuda Index | Day -2 and day 55
  To assess the effect of AZD4076 on Matusda Index
AUC0-24 of AZD4076 and longmer and shortmer metabolites | Dosing day 1 and day 42
  To characterize pharmacokinetics of AZD4076 by area under the curve to 24 hours
Cmax of AZD4076 and longmer and shortmer metabolites | Dosing day 1 and day 42
  To characterize pharmacokinetics of AZD4076 by peak concentration
Tmax of AZD4076 and longmer and shortmer metabolites | Dosing day 1 and day 42
  To characterize pharmacokinetics of AZD4076 by time to peak concentration
CLR of AZD4076 and longmer and shortmer metabolites | Day 1 and 42
  To characterize pharmacokinetics of AZD4076 by clearance
fe% of AZD4076 and longmer and shortmer metabolites | Dosing day 1 and day 42
  To characterize pharmacokinetics of AZD4076 by fraction excreted in urine
Ae of AZD4076 and longmer and shortmer metabolites | Dosing day 1 and day 42
  To characterize pharmacokinetics of AZD4076 by amount excreted in urine

CONTACTS AND LOCATIONS:
Overall Officials: Linda Morrow, MD, Principal Investigator — ProSciento, Inc.